CLINICAL TRIAL: NCT06143982
Title: Effectiveness of a Brief Intensive Trauma Treatment for Adolescents With (Subclinical) PTSD: a Multi-center Randomized Controlled Trial
Brief Title: Effectiveness of a Brief Intensive Trauma Treatment for Adolescents With (s)PTSD: a Multi-center RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. R.J.L. (Ramón) Lindauer, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Effectstudie BITT
Record Dates: First submitted 2023-09-01; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-09

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; Trauma; Intensive treatment; BITT; Adolescents
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A two-arm, mutli-center, randomized controlled trial (RCT). Adolescents (12-18 years old) with (s)PTSD will be randomly allocated by an independent researcher to the intervention group (n=50) versus a waitlist control group (WLCG; n=50), stratified by center. If allocated to the intervention group, participants follow the Brief Intensive Trauma Treatment (BITT). When allocated to the WLCG, participants receive BITT after a 3 months waiting period. Measurements are done at comparable time intervals for both groups: at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intensive Trauma Treatment (Experimental): If allocated to the intervention group, participants follow the Brief Intensive Trauma Treatment (BITT).
  Interventions: Behavioral: Brief Intensive Trauma Treatment
- Waitlist control group (No Intervention): When allocated to the WLCG, participants receive BITT after a 3 months waiting period. The WLCG receives no care during the treatment phase (one week) of the intervention group. Besides this week the WLCG can undergo every treatment including EMDR and TF-CBT during the 3 months waiting period.

INTERVENTIONS:
Behavioral: Brief Intensive Trauma Treatment — BITT is an outpatient, intensive, one-week individual trauma therapy program. BITT is based on well-established protocols, consisting of two 90-minutes trauma therapy sessions a day (trauma exposure in the morning and EMDR in the afternoon), two psychomotor therapy sessions a day (1x60 minutes, 1x45 minutes), one 90-minutes psycho-education and social support skill training for parents a day, and a 90-minutes family therapy session at the end of the week (sharing the trauma narrative).
  Arms: Brief Intensive Trauma Treatment

SUMMARY:
The primary objective of this study is to examine the effectiveness of a Brief Intensive Trauma Treatment (BITT) for adolescents with (s)PTSD.

DETAILED DESCRIPTION:
This study is a multi-center, single-blinded RCT. Adolescents (12-18 years old) with (s)PTSD will be randomly allocated by an independent researcher to the BITT (n=50) versus a waitlist control group (WLCG; n=50), stratified by center. Measurements are done at comparable time intervals for both groups: at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up. The WLCG receives BITT after the 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* 12-18 years of age;
* with a history of psychological trauma (conform the Life Events Checklist of the Clinician Administered PTSD Scale for Children and Adolescents DSM-5 (CAPS-CA DSM-5) (Nader, 2004; van Meijel et al., 2019);
* at least subthreshold PTSD criteria, conform the CAPS-CA DSM-5, i.e.;

  * fully meeting criterion A, F and G and at least one symptom of criteria B, C, D and E;
  * or fully meeting criterion A, F, G and at least the B, C, D or E symptom clusters;
* and written informed consent must be provided by the adolescent and, for adolescents aged 12-15 years, all legal guardians.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study in case of:

* inability to speak and write Dutch;
* estimated or determined mental retardation (IQ <70);
* suffering from ongoing trauma by a parent who is part of the adolescent's current primary-care system.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Posttraumatic stress symptoms (CAPS-CA) | PTSD symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The primary objective of this study is to test the effectiveness of BITT versus a WLCG on adolescents (12-18 years) with (s)PTSD. PTSD symptoms will be assessed by the Clinician Administered PTSD Scale for Children and Adolescents DSM-5 (CAPS-CA DSM 5; Van Meijel et al., 2013). Additionally, the effectiveness of BITT versus regular trauma treatment (i.e., TF-CBT and EMDR) on (s)PTSD symptoms will be tested.
Changes in Posttraumatic stress symptoms (KJTS) | PTSD symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The primary objective of this study is to test the effectiveness of BITT versus a WLCG on adolescents (12-18 years) with (s)PTSD. PTSD symptoms will be assessed by the Child and Adolescent Trauma Screening (In Dutch: Kind en Jeugd Trauma Screener (KJTS; Kooij & Lindauer, 2019). Additionally, the effectiveness of BITT versus regular trauma treatment (i.e., TF-CBT and EMDR) on (s)PTSD symptoms will be tested.

SECONDARY OUTCOMES:
Changes in Anger symptoms (PROMIS) | Anger symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The second objective is to test the effectiveness of BITT versus a WLCG on anger symptoms. Anger symptoms will be measures with the Patient-Reported Outcomes Measurement Information System (PROMIS; Terwee et al., 2014). Additionally, the effectiveness of BITT versus regular trauma treatment (i.e., TF-CBT and EMDR) on anger will be tested.
Changes in Anger symptoms (SCID-5 Junior) | Anger symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  Anger symptoms will also be measures with the Structured Clinical Interview for DSM-5 Childhood Disorders (SCID-5 Junior; module 12 Disruptive, impulse control and other behavioral disorders; Wante et al., 2020). The SCID-5 module will be administered when the adolescent scores T ≥ 60 on the PROMIS questionnaire.
Changes in Anxiety symptoms (PROMIS) | Anxiety symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The third objective is to test the effectiveness of BITT versus a WLCG on anxiety symptoms. Anxiety symptoms will be measures with the Patient-Reported Outcomes Measurement Information System (PROMIS; Terwee et al., 2014). Additionally, the effectiveness of BITT versus regular trauma treatment (i.e., TF-CBT and EMDR) on anxiety will be tested.
Changes in Anxiety symptoms (SCID-5-Junior) | Anxiety symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  Anxiety symptoms will also be measures with the Structured Clinical Interview for DSM-5 Childhood Disorders (SCID-5 Junior; Module 6 Anxiety disorder; Wante et al., 2020). The SCID-5 module will be administered when the adolescent scores T ≥ 60 on the PROMIS questionnaire.
Changes in Depression symptoms (PROMIS) | Depression symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The fourth objective is to test the effectiveness of BITT versus a WLCG on depression symptoms. Depression symptoms will be measures with the Patient-Reported Outcomes Measurement Information System (PROMIS; Terwee et al., 2014). Additionally, the effectiveness of BITT versus regular trauma treatment (i.e., TF-CBT and EMDR) depression symptoms will be tested.
Changes in Depression symptoms (SCID-5-Junior) | Depression symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  Depression symptoms will also be measures with the Structured Clinical Interview for DSM-5 Childhood Disorders (SCID-5 Junior; Module 3 Depressive mood disorders; Wante et al., 2020). The SCID-5 module will be administered when the adolescent scores T ≥ 60 on the PROMIS questionnaire.
Changes in Quality of life | Quality of life is measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The fifth objective of this study is to examine the effectiveness of BITT versus a WLCG on quality of life. Quality of life will be measures with the EuroQol-5D (EuroQol-Group, 2009). Additionally, the effectiveness of BITT versus regular trauma treatment (i.e., TF-CBT and EMDR) on quality of life will be tested.
Changes in Risk-behavior and safety | Risk-behavior and safety is measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The sixth objective is to test if BITT is a safe intervention. This will be measured with a risk-behavior and safety questionnaire based on previous work by Hendriks et al. (2017) regarding: self-harm, suicidality and aggressive behavior.
Dropout rates | Dropout is measures at each day of the BITT week (in total 5 days).
  The seventh objective is to examine if BITT leads to less drop out rates. Drop outs will be documented in an Excel file (yes/no).
Cost-effectiveness | Cost-effectiveness is measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  The eighth objective is to examine the cost-effectiveness of BITT. Cost-effectiveness will be measured with the Treatment Inventory of Costs in Psychiatric clients (TiC-PY/proxy) (Bouwmans et al., 2012).

OTHER OUTCOMES:
Age (moderator) | Age is documented at pre-treatment (T0).
  Age will be studied as a moderator on the effectiveness of BITT on PTSD.
Sex (moderator) | Sex is documented at pre-treatment (T0).
  Sex will be studied as a moderator on the effectiveness of BITT on PTSD.
Socioeconomic status (SES; moderator) | SES is documented at pre-treatment (T0).
  SES will be studied as a moderator on the effectiveness of BITT on PTSD.
Type of trauma (moderator) | Type of trauma is measured at pre-treatment (T0).
  Type of trauma will be studied as a moderator on the effectiveness of BITT on PTSD. Type of trauma will be assessed with de CAPS-CA DSM-5 (Van Meijel et al., 2013).
Number of traumatic events (moderator) | Number of traumatic events is measured at pre-treatment (T0).
  Number of traumatic events will be studied as a moderator on the effectiveness of BITT on PTSD. Number of traumatic events will be assessed with the CAPS-CA DSM-5 (Van Meijel et al., 2013).
Comorbidity (anger symptoms; moderator) | Anger symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  Comorbidity (anger symptoms; moderator) will be studied as moderator on the effectiveness of BITT on PTSD. Anger will be assessed with the PROMIS (Terwee et al., 2014).
Comorbidity (anxiety symptoms moderator) | Anxiety symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  Comorbidity (anxiety symptoms; moderator) will be studied as moderator on the effectiveness of BITT on PTSD. Anxiety symptoms will be assessed with the PROMIS (Terwee et al., 2014).
Comorbidity (depression symptoms; moderator) | Depression symptoms are measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  Comorbidity (depression symptoms; moderator) will be studied as moderator on the effectiveness of BITT on PTSD. Depression symptoms will be assessed with the PROMIS (Terwee et al., 2014).
Parental PTSD (moderator) | Parental PTSD is measured at pre-treatment (T0), directly after BITT or WLCG (T1) and at 3 (T2), 6 (T3) and 9 (T4) months follow-up.
  Parental PTSD will be studied as a moderator on the effectiveness of BITT on PTSD. Parental PTSD will be assessed with the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) (Blevins et al., 2015).
Treatment center (Participating centers: Levvel/Karakter/Mental Health Caribbean; moderator) | Treatment center (Levvel, Karakter, Mental Health Caribbean) is documented at pre-treatment (T0).
  Treatment center (Levvel, Karakter, Mental Health Caribbean) will be studied as a moderator on the effectiveness of BITT on PTSD.
Residency (urban/rural; moderator) | Residency is documented at pre-treatment (T0).
  Residency (urban/rural) will be studied as a moderator on BITT dropout.
Ethnicity | Ethnicity is documented at pre-treatment (T0).
  Ethnicity will be studied as a moderator on BITT dropout.

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Lindauer, Prof. dr., Principal Investigator — Amsterdam UMC, location AMC/Levvel
Locations (3):
- Mental Health Caribbean, Kralendijk, Bonaire, Saint Eustatius and Saba
- Netherlands (2):
  - Amsterdam UMC, location AMC/Levvel, Amsterdam, North Holland
  - Karakter, Almelo, Overijsel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Westerveld MM, van der Mheen M, Knipschild R, Maijer K, de Keizer-Altink ME, Albisser N, Hoekstra MJE, Timmermans-Jansen A, Zijp R, Krabbendam AA, van Steensel FJAB, Kan KJ, Huyser C, Staal WG, Utens EMWJ, Lindauer RJL. Short- and Long-Term Effectiveness of Brief Intensive Trauma Treatment for Adolescents With Posttraumatic Stress Disorder and Their Caregivers: Protocol for a Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 30;14:e66115. doi: 10.2196/66115. PMID 40306642